CLINICAL TRIAL: NCT01600950
Title: Pharmacodynamics of LY2963016 Compared to LANTUS® in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Study to Compare LY2963016 to Lantus After a Single Dose to Participants With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 13831; I4L-MC-ABEE (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — LY2963016 insulin glargine; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2963016 (Experimental): A single 0.3 units per kilogram (U/kg) dose of LY2963016 will be administered subcutaneously followed by a minimum washout period of 7 days.
  Interventions: Drug: LY2963016
- Lantus (Active Comparator): A single 0.3 U/kg dose of Lantus will be administered subcutaneously followed by a minimum washout period of 7 days.
  Interventions: Drug: Lantus

INTERVENTIONS:
Drug: LY2963016 — Single 0.3 U/kg dose administered subcutaneously
  Arms: LY2963016
Drug: Lantus — Single 0.3 U/kg dose administered subcutaneously
  Arms: Lantus

SUMMARY:
The study involves a single injection of LY2963016 and a single injection of Lantus, on 2 separate occasions in participants with type I diabetes. Following each dose, participants will undergo a glucose clamp which lasts for 42 hours each time. There will be at least 7 days between the two periods, during which time there will be no study treatment, but participants will resume their regular therapy. The duration of this study can be up to 9.5 weeks. The purposes of this study are to understand how the blood sugar lowering effect of LY2963016 compares to that of Lantus, and to determine how LY2963016 and Lantus are metabolized by participants with type I diabetes.

ELIGIBILITY:
Inclusion Criteria:

* have type 1 diabetes mellitus (T1DM) based on the disease diagnostic criteria
* have had a duration of diabetes ≥1 year
* have hemoglobin A1c ≤10.0%
* have fasting C-peptide ≤0.3 nanomoles per liter (nmol/L)
* have a body mass index ≤29 kilograms per square meter (kg/m²)
* have venous access sufficient to allow blood sampling and cannulation for clamp procedures

Exclusion Criteria:

* are currently enrolled in, have completed, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device
* have a total insulin requirement >1.2 units per kilogram per day (U/kg/day)
* have a history of proliferative retinopathy
* have known allergies to insulin glargine, insulin lispro, heparin, or related compounds
* have an electrocardiogram (ECG) reading considered outside the normal limits
* have an abnormal blood pressure
* have abnormal clinical laboratory tests
* have a history or presence of/significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs
* history of deep leg vein thrombosis or a frequent appearance of deep leg vein thrombosis in first-degree relatives
* show evidence of significant active neuropsychiatric disease
* regular use of known drugs of abuse and/or show positive findings on drug screening
* show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies
* show evidence of hepatitis C and/or positive hepatitis C antibody
* show evidence of hepatitis B and/or positive hepatitis B surface antigen
* are women with a positive pregnancy test or women who are lactating
* have an average weekly alcohol intake that exceeds 21 units per week (males) or 14 units per week (females)
* had more than 1 episode of severe hypoglycemia within 6 months prior to study
* undergoing therapy for a malignancy other than basal cell or squamous cell skin cancer
* had a blood transfusion or severe blood loss within 3 months; made a blood donation within 30 days prior to study entry; or have known hemoglobinopathy, haemolytic anemia, or sickle cell anemia
* are receiving systemic glucocorticoid therapy
* have irregular sleep/wake cycle (for example, participants who sleep during the day and work during the night)
* show a history of adverse reactions to heparin, including heparin-induced thrombocytopenia
* smoke more than 10 cigarettes (or equivalent other tobacco products) per day

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neuss, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomized, 2-period, 2-sequence, crossover study.
Groups:
- LY2963016/Lantus: A single 0.3 units per kilogram (U/kg) dose of LY2963016 was administered subcutaneously on Day 1 during Period 1 followed by a minimum washout period of 7 days.
  A single 0.3 U/kg dose of Lantus was administered subcutaneously on Day 1 during Period 2.
- Lantus/LY2963016: A single 0.3 U/kg dose of Lantus was administered subcutaneously on Day 1 during Period 1 followed by a minimum washout period of 7 days.
  A single 0.3 U/kg dose of LY2963016 was administered subcutaneously on Day 1 during Period 2.
Period: Period 1
Arm/Group | LY2963016/Lantus | Lantus/LY2963016
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Period 2
Arm/Group | LY2963016/Lantus | Lantus/LY2963016
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- All Participants: A single 0.3 units/kilogram (U/kg) dose of either LY2963016 or LANTUS was administered subcutaneously on Day 1 of Periods 1 or 2.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 20

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamics: Duration of Action of LY2963016 and Lantus
Description: Duration of action is defined as the period of time elapsed between dose administration and the time at which the participant's blood glucose is consistently >150 milligrams/deciliter (mg/dL) without any glucose infusion. Participants whose blood glucose did not rise to 150 mg/dL were censored 42 hours postdose.
Time Frame: Periods 1 and 2: Baseline up to 42 hours postdose
Population: All randomized participants who received study drug during Periods 1 or 2. Participants were analyzed based on treatment they received. The numbers of participants censored were 7 for both LY2963016 and Lantus groups. Maximum duration of actions is based on participants who reached the end of action before 42 hours: 13 participants for both groups.
Measure: Median (Full Range); unit: hours (hr)
Groups:
- LY2963016: A single 0.3 units per kilogram (U/kg) dose of LY2963016 was administered subcutaneously on Day 1 of Periods 1 or 2.
- Lantus: A single 0.3 U/kg dose of Lantus was administered subcutaneously on Day 1 of Periods 1 or 2.
Arm/Group | LY2963016 | Lantus
Number analyzed (Participants) | 20 | 20
hours (hr) | 37.13 [2.8 to 40.5] | 40.00 [2.0 to 41.5]

2. Secondary Outcome: Maximum Glucose Infusion Rate (Rmax)
Description: Rmax is the maximum infusion rate of glucose administered intravenously needed to maintain a target blood glucose level of 100 milligrams/deciliter (mg/dL) [5.6 millimoles/Liter (mmol/L)] and is used to measure the study drug action over time as measured by the euglycaemic clamp procedure. During the euglycaemic clamp procedure, blood glucose concentrations are held constant after the administration of study drug by adjusting the exogenous glucose infusion rate. Data presented are the maximum infusion rates, adjusted by body weight.
Time Frame: Periods 1 and 2: Baseline up to 42 hours postdose
Population: All randomized participants who received the study drug during Periods 1 or 2. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams/kilogram/minute (mg/kg/min)
Arm/Group | LY2963016 | Lantus
Number analyzed (Participants) | 20 | 20
milligrams/kilogram/minute (mg/kg/min) | 0.530 (254) | 0.611 (310)

3. Secondary Outcome: Total Glucose Infused (Gtot)
Description: Gtot is the total glucose infusion over the clamp duration and is used to measure the study drug action over time as measured by the euglycaemic clamp procedure. During the euglycaemic clamp procedure, blood glucose concentrations are held constant after the administration of study drug by adjusting the exogenous glucose infusion rate. Data presented are the total glucose infused, adjusted by body weight.
Time Frame: Periods 1 and 2: Baseline up to 42 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams/kilogram (mg/kg)
Arm/Group | LY2963016 | Lantus
Number analyzed (Participants) | 20 | 20
milligrams/kilogram (mg/kg) | 4.60 (1090) | 6.52 (1160)

4. Secondary Outcome: Time of Maximum Glucose Infusion Rate (tRmax)
Description: tRmax is the time to reach maximum glucose infusion rate and is used to measure the study drug action over time as measured by the euglycaemic clamp procedure. During the euglycaemic clamp procedure, blood glucose concentrations are held constant after the administration of study drug by adjusting the exogenous glucose infusion rate.
Time Frame: Periods 1 and 2: Baseline up to 42 hours postdose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | LY2963016 | Lantus
Number analyzed (Participants) | 20 | 20
hours (hr) | 9.90 [1.50 to 30.1] | 11.7 [1.00 to 29.6]

5. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY2963016 and Lantus
Description: Cmax was not analyzed because of insufficient data due to concentrations being below the quantifiable lower limit of the assay.
Time Frame: Periods 1 and 2: Baseline up to 42 hours postdose
Population: No participants were analyzed because of insufficient data.
Arm/Group | LY2963016 | Lantus
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-time Curve (AUC) of LY2963016 and Lantus
Description: AUC was not analyzed because of insufficient data due to concentrations being below the quantifiable lower limit of the assay.
Time Frame: Periods 1 and 2: Baseline up to 42 hours postdose
Population: No participants were analyzed because of insufficient data.
Arm/Group | LY2963016 | Lantus
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | LY2963016 | Lantus
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/20 | 3/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2963016 (N=20) | Lantus (N=20)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days